CLINICAL TRIAL: NCT07330648
Title: Evaluation of the Efficacy and Safety of Crisugabalin Capsules Versus Placebo and Venlafaxine Extended-Release (XR) Capsules in Chinese Patients With Generalized Anxiety Disorder: A Prospective, Multicenter, Randomized, Double-Blind, Double-Dummy, Active- and Placebo-Controlled Clinical Trial.
Brief Title: Prospective Clinical Trial of Crisugabalin Capsules in the Treatment of Generalized Anxiety Disorder
Acronym: CEASE-GAD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, The First Affiliated Hospital of Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK16149-502
Record Dates: First submitted 2025-11-24; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-10

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — BID protein, human; tebufenozide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crisugabalin 80mg/day group (Experimental): Crisugabalin 20mg, orally twice a day; treatment period: 8 weeks fixed dose. Open-label extension phase: Crisugabalin 40mg, orally twice a day; treatment period: 4 weeks fixed dose.
  Interventions: Drug: Crisugabalin 20mg bid
- Venlafaxine Extended-Release (XR) Capsules 150mg/day group (Experimental): Drug: Venlafaxine-XR 75mg bid Venlafaxine-XR 75mg, orally once a day and the second dose of placebo was administered; treatment period: 8 weeks fixed dose.
  Interventions: Drug: Venlafaxine-XR 75mg bid
- Placebo-Control group (Placebo Comparator): Drug: Crisugabalin capsules mimic 0mg/capsule bid Crisugabalin capsules mimic 0mg/capsule, orally twice a day; treatment period: 8 weeks fixed dose.
  Drug: Venlafaxine-XR capsules mimic, 0mg/capsule, bid Venlafaxine-XR capsules mimic, 0mg/capsule, orally twice a day; treatment period: 8 weeks fixed dose.
  Interventions: Drug: Crisugabalin capsules mimic 0mg/capsule bid

INTERVENTIONS:
Drug: Crisugabalin 20mg bid — Crisugabalin 20mg bid Crisugabalin 20mg, orally twice a day; treatment period: 8 weeks fixed dose. Open-label extension phase: Crisugabalin 40mg, orally twice a day; treatment period: 4 weeks fixed dose.
  Other Names: HSK16149
  Arms: Crisugabalin 80mg/day group
Drug: Venlafaxine-XR 75mg bid — Venlafaxine-XR 75mg bid Venlafaxine-XR 75mg, orally once a day and the second dose of placebo was administered; treatment period: 8 weeks fixed dose.
  Other Names: Venlafaxine-XR
  Arms: Venlafaxine Extended-Release (XR) Capsules 150mg/day group
Drug: Crisugabalin capsules mimic 0mg/capsule bid — Crisugabalin capsules mimic 0mg/capsule, orally twice a day; treatment period: 8 weeks fixed dose.
  Drug: Venlafaxine-XR capsules mimic, 0mg/capsule, bid Drug: Venlafaxine-XR capsules mimic, 0mg/capsule, bid Venlafaxine-XR capsules mimic, 0mg/capsule, orally twice a day; treatment period: 8 weeks fixed dose.
  Other Names: Crisugabalin capsules mimic; Venlafaxine-XR capsules mimic
  Arms: Placebo-Control group

SUMMARY:
A placebo-controlled superiority design was used to evaluate the efficacy of 40 mg/ day of Crisugabalin capsules in the treatment of GAD.

DETAILED DESCRIPTION:
This was a prospective, multicenter, randomized, double-blind, double-dummy, active- and placebo-controlled clinical trial.

Qualified subjects, according to the ratio of 1:1:1, were randomized into Crisugabalin group, Venlafaxine-control group and placebo-control group, and received a double-blind treatment course of 8 weeks. After completing the 8-week double-blind treatment period, subjects will officially conclude the study or voluntarily enter a 4-week open-label extension treatment phase. During the open-label extension phase, all subjects will receive Crisugabalin 80 mg/day (40 mg bid). Participants were followed from baseline outpatient visit until end of the follow-up period (14 weeks and 9 visits in total).

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily participate in the trial, and provide written informed consent form (ICF);
* Male or female aged ≥18 years (inclusive of the threshold value);
* Met the diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for generalized anxiety disorder (GAD) and confirmed by the Brief International Neuropsychiatric Interview (M.I.N.I.);
* Require pharmacological treatment for psychiatric symptoms;
* Hamilton Anxiety Scale (HAMA) score ≥20, Hamilton Depression Scale (HAMD-17) score ≤2, Clinical Global Impression Scale (CGI-S) score ≥4 at screening and baseline Points;

Exclusion Criteria:

* subjects with serious suicide risk at present, or HAMD-17 item 3-suicide score ≥3;
* subjects with HAMD-17 > 17;
* subjects whose HAMA scores decreased by ≥20% in the baseline period compared with the screening period:
* Those who met the DSM-5 diagnostic criteria for other mental disorders except GAD;
* subjects with previous history of depression, obsessive-compulsive disorder, bipolar disorder, psychotic disorder, factitious disorder and somatoform disorder; There were severe personality disorders, especially antisocial, borderline, or histrionic personality disorder, which were judged by the investigator to affect the patient's adherence to the study protocol;
* Alcohol or drug abuse or dependence within 180 days before screening;
* With severe or unstable has clinical significance of somatic disease, including any cardiovascular, cancer, kidney, respiratory, endocrine (including abnormal thyroid function), digestion, blood (such as with bleeding tendency) or nervous system diseases;
* History of inadequate response to at least two prior antidepressant drugs and/or benzodiazepines after adequate dose and duration of treatment (i.e., at least 4 weeks at a clinically appropriate dose), or failure to achieve sufficient clinical efficacy with pregabalin ≥300 mg/day (i.e., subject-reported insufficient response or lack of meaningful clinical improvement).
* History of severe hypersensitivity reactions (e.g., anaphylaxis) or allergies to at least two classes of drugs (including photosensitivity), or known hypersensitivity to pregabalin, the investigational drug, structurally related compounds, or any of their excipients.
* subjects whose physical examination or vital signs were abnormal and clinically significant (e.g. inadequately controlled hypertension, systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg);
* subjects with a history of epilepsy or any other disease that may induce seizures, except convulsions caused by febrile convulsions in children;
* Severe hematologic, hepatic or renal dysfunction during the screening period, the subject will be excluded if: a. Neutrophils < 1.5 × 10^9/L, or platelet < 90 × 10^9/L, or hemoglobin < 100 g/L; b. AST/ALT > 2.5 × upper limit of normal (ULN), or TBIL > 1.5 × ULN; c. Estimation of glomerular filtration rate (eGFR) < 60 mL/min / 1.73 m^2; d. Creatine kinase > 2.0 × ULN.
* Clinically significant abnormalities on electrocardiography (QT interval corrected by Fridericia method: ≥450 ms for men or ≥470 ms for women) or conditions deemed ineligible by the investigators;
* Subjects who had undergone psychiatric surgery, electroconvulsive therapy or transcranial magnetic stimulation within 90 days before screening;
* Use of β-blockers within 90 days prior to screening with an ongoing need for continued treatment;
* Receiving systemic psychotherapy or other non-pharmacological treatments (e.g., acupuncture, hypnosis, or phototherapy) within 6 weeks before the baseline visit;
* Subjects with dysphagia or inability to tolerate oral medications.
* Subjects with active gastrointestinal disorders (including any history of gastrointestinal surgery) that, in the investigator's judgment, may interfere with the absorption of the investigational drug.
* Those who had used benzodiazepines within -7 to -1 days before screening, such as lorazepam, oxazepam, and alprazolam for less than 5 half-lives; The use of benzodiazepines with longer half-lives, such as diazepam, clonazepam, nitrazepam, estazolam, and flurazepam, not more than 5 half-lives or less than 30 days from the screening period, or the use of barbiturates not more than 5 half-lives or less than 30 days from the screening period;
* Patients who discontinued traditional Chinese medicine, melatonin, and St. John's wort for less than 3 days before the baseline visit;
* Pregnant or preparing for pregnancy or breastfeeding during the study period, or subjects were not willing to use reliable contraceptives methods from the date of ICF signature until 28 days after the last trial drug administration, or planning to use progesterone contraceptives during this period;
* Individuals engaged in potentially hazardous mechanical operations such as working at heights or operating motor vehicles.
* Participants enrolled in other clinical trials within 30 days before screening;
* Subjects with other conditions deemed by the investigator to be ineligible for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Anxiety (HAMA) scale score after 8 week treatment | from baseline to week 8
  The Hamilton Anxiety (HAMA) scale score reflects the severity of the subjects anxiety symptoms. The primary efficacy end point was the change from baseline to week 8 in HAMA total score to determine the superiority of crisugabalin capsules over placebo. The larger the difference between crisugabalin capsules over placebo, the better the curative effect.The HAMA consists of 14 items that encompass both psychological and somatic symptoms of anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.

SECONDARY OUTCOMES:
Change in Hamilton anxiety scale score after treatment | from baseline to week 8
  One of the secondary efficacy end point was the change from baseline to week 8 in Hamilton anxiety scale to determine the superiority of crisugabalin capsules over placebo. The larger the difference between crisugabalin capsules over placebo, the better the curative effect.The HAMA consists of 14 items that encompass both psychological and somatic symptoms of anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Change in each factor score and item score of Hamilton anxiety scale | from baseline to week 8
  One of the secondary efficacy end point was the change from baseline to week 8 in each factor score and item score of Hamilton anxiety scale to determine the superiority of crisugabalin capsules over placebo. The larger the difference between crisugabalin capsules over placebo, the better the curative effect. The HAMA consists of 14 items that encompass both psychological and somatic symptoms of anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Clinical global impression of improvement score | the end of week 4 and 8
  Subjective improvement of crisugabalin capsules will be assessed using Clinical Global Impression of Improvement (CGI-I) score at week 4 and 8. The larger the difference between crisugabalin capsules over placebo, the better the curative effect. The CGI-I scale is used to measure the clinician's assessment of how much the participant's illness has improved or worsened relative to baseline. The CGI-I comprises one item with 7 possible ratings (1-7 points), where a lower score indicates improvement, and a higher score indicates worsening.
Clinical global impression of severity score | the end of week 4 and 8
  Subjective severity of crisugabalin capsules will be assessed by the change from baseline to week 4 and 8 with Clinical global impression of severity (CGI-S) score, to determine the superiority of crisugabalin capsules over placebo. The larger the difference between crisugabalin capsules over placebo, the better the curative effect. The CGI-S scale assesses the clinician's impression of the participant's current severity of illness relative to the clinician's experience with patients who have the same diagnosis. The CGI-S comprises one item with 7 possible ratings (1-7 points), where a higher score indicates more severe illness.
Complete remission rate | the end of week 8
  Complete remission rate was the proportion of subjects with HAMA total scale score ≤7 at the end of week 8. The larger the difference between crisugabalin capsules over placebo, the better the curative effect. The HAMA consists of 14 items that encompass both psychological and somatic symptoms of anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Response rate | the end of week 8
  Response rate was the proportion of subjects with HAMA total score decreased by ≥50% from baseline to week 8. The larger the difference between crisugabalin capsules over placebo, the better the curative effect. The HAMA consists of 14 items that encompass both psychological and somatic symptoms of anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Rapid-onset rate | the end of week 1 and 2
  Rapid-onset rate was the proportion of subjects with HAMA total score decreased by ≥20% from baseline to week 1 and 2. The larger the difference between crisugabalin capsules over placebo, the better the curative effect. The HAMA consists of 14 items that encompass both psychological and somatic symptoms of anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.

OTHER OUTCOMES:
Exploratory Analysis | Form baseline to week 8
  A descriptive statistical analysis will be performed to evaluate the change from baseline in HAMA total score for Venlafaxine-XR.
  The HAMA consists of 14 items that encompass both psychological and somatic symptoms of anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Adverse events (AEs） | Form baseline to week 8
  number and severity of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No